CLINICAL TRIAL: NCT05226312
Title: The Effect of Warm Wet Application in the Care of Peripheral Intravenous Catheter-related Phlebitis.
Brief Title: Phlebitis Care and Warm Wet Application
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Ordu University (Other)
Responsible Party: Principal Investigator, Fatma Aksoy, Research Assistant, Ordu University
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Supportive Care
Other Study IDs: OrduSBF
Record Dates: First submitted 2021-10-28; First posted 2022-02-07 (Actual); Last update posted 2022-09-09 (Actual); Status verified 2022-09

CONDITIONS: Pain; Phlebitis; Nursing Caries
Keywords: Pain; quality of health care; Peripheral Intravenous Catheter
MeSH Terms: conditions — Pain; Phlebitis

STUDY DESIGN:
Intervention Model Description: Randomize Control experimental study
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Local Warm Compress (Experimental): They are gauze covers brought to a certain temperature (temperature varies between 26-34°C or 79-93°F in warm applications) as a compress material, or wraps and covers that can be reheated.
  Interventions: Other: Local Warm Compress
- Not Local Warm Compress (No Intervention): No warm wet application will be made to this group. It will be tracked for only 3 days.

INTERVENTIONS:
Other: Local Warm Compress — The warm application will be made by the researcher for 15 minutes three times a day according to the local warm application process steps.
  Arms: Local Warm Compress

SUMMARY:
Phlebitis is an inflammation of the tunica intima layer of the vein. Intravenous administration of drugs with high pH and osmolarity via a peripheral intravenous catheter damages the vascular structure, causing the drug to leak out of the vessel and cause phlebitis. Planning the care of the area where phlebitis occurs is the responsibility of the nurses. When phlebitis symptoms are seen, the infusion is terminated, the treatment is continued from another area, the extremity is elevated, and warm application is started. However, studies in the literature on what, how many degrees, how many times a day, and how long the warm application should be made are limited. Therefore, this planned thesis study was designed as a randomized controlled experimental study to determine the effect of warm wet application in the care of peripheral intravenous catheter-related phlebitis. The study will be carried out in Ordu University Training and Research Hospital oncology, hematology, palliative, infection, and obstetrics services. The population of the study will be the patients with phlebitis symptoms, and the sample will be 70 patients determined by G power analysis. Volunteer patients with phlebitis symptoms after drug infusion with a peripheral intravenous catheter will be included in the study. Data will be obtained using the "Patient Information Form", "Phlebitis Follow-up Form" and "Phlebitis Care Schedule". The patients included in the study will be divided into experimental and control groups by the randomization method. A warm wet compress will be applied to the phlebitis developing area of the patients in the experimental group, three times a day for three days. No intervention will be made in the control group. The data will be evaluated by using the SPSS 22.0 package program at a significance level of p<0.05 with a 95% confidence interval, and by Student-t or Mann-Whitney-U test in independent groups according to their suitability for normal distribution. It is thought that the results of the study will reduce the symptoms of phlebitis, guide nurses towards care and increase patient satisfaction.

DETAILED DESCRIPTION:
Peripheral intravenous (PIV) therapy is the process of injecting fluid directly into the patient's vein. In cases where fluid and electrolyte balance cannot be achieved in patients who cannot be fed orally, in the administration of chemotherapy, antibiotics, and other intravenously administered drugs, intravenous therapy is frequently used in patients followed at the intensive care level, and fluids are given directly into the bloodstream. Although peripheral IV therapy has many benefits on the patient, complications such as phlebitis, infiltration, extravasation, thrombosis, cellulitis, and bloodstream infection may occur. The occurrence of these complications is related to inadequate catheter care, length and diameter of the catheter, length of stay in the vein, the substance it is produced, the patient's vascular structure and position, the type and flow rate of the given fluid, the length of stay in the hospital, and the individual characteristics of the patient.

Peripheral intravenous catheter complications may develop during catheterization or during infusion or may occur 24-96 hours after catheter removal. When these complications are encountered, the duration of the hospital stay of the patient is prolonged, and as a result, mortality and morbidity rates increase. The incidence of PIV catheter complications in our country is close to 50%. Among the complications, the most common and the most important complication is phlebitis. While the incidence of phlebitis is between 24.3% and 31.8% according to national studies, this rate is between 2.63% and 44% in international studies. Studies have reported that the incidence of phlebitis is higher in individuals receiving chemotherapy. Because chemotherapy treatments are usually administered by the PIV route. The irritant, vesicant, non-vesicant properties of chemotherapy drugs, high pH and osmolarity levels, and repeated cure treatments damage peripheral veins. In addition, antibiotics, hypertonic solutions, blood, and nutritional products, and analgesics are risk factors for the development of phlebitis.

Phlebitis is defined as the inflammation of the tunica intima layer of the vein. Phlebitis occurs in three ways: mechanical, chemical, and bacterial. Mechanical phlebitis; It is seen for reasons such as the individual characteristics of the patient, the catheter insertion site, the catheter type, and number, the material used in the catheter fixation, the length of time the catheter stays in the vein, the treatment time, the skill of the person inserting the catheter, the determination of the appropriate vein, the fluid flow rate, the use of infusion pumps, and the number of drugs given. Chemical phlebitis; It is seen when irritating drugs are given intravenously in a liquid with a density of 600 mOsm/lt or the pH of the fluids is less than 5 and greater than 9. Bacterial phlebitis is caused by factors such as cleaning the area with antiseptic, the frequency of changing the infusion set from the material on which the catheter is fixed, and the care of the catheter site. Symptoms of phlebitis are redness, erythema, pain, edema, palpable stiffness along the vein (venous cord), prominence of the venous line, tenderness, discharge, and warmth. The catheter site should be followed up with the "Visual Infusion Phlebitis Diagnostic Scale" in terms of these symptoms. However, in a study conducted by Arpa and Cengiz, it was found that nurses did not know the scale and had a lack of knowledge. Therefore, not following the catheter site and not recognizing the symptoms increase the incidence of phlebitis. When one of the symptoms of phlebitis is observed, the degree of phlebitis should be defined according to the scale and appropriate nursing interventions should be planned.

In the care of the patient with phlebitis, the infusion should be terminated, the catheter should be removed, the extremity should be elevated, and a new catheter should be inserted to continue treatment from another site. The area where phlebitis develops should not be used for a new catheterization for at least 48 hours. Symptoms such as redness, pain, swelling, and length of venous cord-shaped hardening in the area where phlebitis develops should be followed according to the visual phlebitis scale. In addition, it is stated in the literature that local warm application can be applied to the area with phlebitis symptoms. However, there is no clear information in the literature regarding when to start local warm application, its duration, and frequency.

Local warm application is frequently used by nurses to provide dilatation of blood vessels, to reduce inflammation by increasing oxygen circulation in hypoxic conditions, and for the non-pharmacological treatment of pain and tenderness. Hot/cold applications can be applied in two ways, wet or dry. The web application provides a moist environment in the area, increases blood flow to the area, carries nutrients, leukocytes, and antibodies, and increases the rate of wound healing. Wet application is more effective than dry application as the heat spreads rapidly to the deep tissues. However, changing the compresses frequently is important for the effectiveness of the application, as it causes evaporation with vasodilation and cooling of the skin.

Thermophore, aquathermic pad, hot or cold gel, hot water bath, ice accumulators, electric heating pad, and compresses are used for hot or cold applications. In the research to be conducted, a warm wet compress will be used. Compresses are used to apply local heat. Compress temperature is brought to the range of 26-34°C (79-93°F) for warm application. Compresses can be prepared in a wide variety of sizes and allowed to apply a certain temperature to the body area.

In the literature, it is stated in the literature that in the case of phlebitis, applying warm wet compresses to the affected area can be used to accelerate the blood flow and to reduce sensitivity and pain with the effect of tissue healing in the area. However, studies on this subject are limited. In a study conducted by Annisa et al. (2017) in 36 individuals aged 1 month to 17 years who developed phlebitis, one group was treated with warm water (n=16) and the other group (n=16) with 0.9% NaCl 3 to 4 times a day. Compress was applied for 20 minutes. When the phlebitis area was followed 24 and 48 hours later, it was stated that the degree of phlebitis decreased statistically significantly. In a study conducted by Hidayah et al. (2017) on 40 individuals aged 17-44 years, it was reported that there was a statistically significant difference in vessel diameter before and after warm wet application and reduced phlebitis. In the study of Gauttan and Vati (2016) with 60 individuals, it was found that wet heat and cold application for 20 minutes every two hours is equally effective and can be used for the treatment of phlebitis.

The Infusion Nurses Association (IHD) stated that it is very important to reduce the incidence of phlebitis to 5% and below, to prevent its occurrence, to be recognized early and to take necessary precautions, or to care about it occurs. Nurses working in clinics such as oncology, hematology, and palliative where phlebitis is common should have sufficient knowledge of phlebitis prevention, care, treatment, and practice. Nursing care provided by following current developments and using evidence-based nursing practices will decrease the incidence of phlebitis and increase the quality of care. In the literature, it is stated that warm application can be used in the care of phlebitis. However, it is not specified what the application will be done with, the temperature and how many times a day it will be done. Therefore, the aim of this study is to determine the effect of warm wet application in the care of peripheral venous catheter-related phlebitis.

ELIGIBILITY:
Inclusion Criteria:

* Patients aged 18 and over,
* Taking the medication with a peripheral intravenous catheter,
* Those with phlebitis symptoms and phlebitis symptoms are regularly monitored,
* No application other than extremity elevation after phlebitis was detected,
* Those who are conscious and able to respond

Exclusion Criteria:

* Neutropenia,
* Heat allergy,
* Peripheral vascular disease,
* Having a dialysis catheter in the application area,
* Receiving anticoagulant therapy,
* Those who have an open wound, scar tissue, metal prosthesis in the area where phlebitis develops,
* Unconscious and unresponsive patients discharged,
* Patients wishing to withdraw from the study

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 70 (Actual)
Dates: Start 2022-02-08 (Actual); Primary Completion 2022-03-10 (Actual); Study Completion 2022-04-10 (Actual)

PRIMARY OUTCOMES:
The effect of warm wet application on pain in the care of peripheral intravenous catheter-related phlebitis | approximately 69 days until 10 April 2022
  The degree of pain before and after the application will be evaluated with the Numeric Rating Scale (NRS). Numeric Rating Scale (NRS) takes values between 0 and 10 points. As the pain score increases, the pain level also increases. Patients included in the study will be evaluated for approximately 69 days until April 10, 2022.
The effect of hot wet application on redness in the care of peripheral intravenous catheter-related phlebitis. | approximately 69 days until 10 April 2022
  The degree of redness will be determined with Opsite Flexigirit before and after application. After the warm wet application, the degree of redness will be determined again and the effectiveness of the warm wet application will be evaluated. Patients included in the study will be evaluated for approximately 69 days until April 10, 2022.
The effect of warm wet application on edema in the care of peripheral intravenous catheter-related phlebitis | approximately 69 days until 10 April 2022
  Before and after the warm wet application, the extent of edema will be determined with Opsite Flexigirit. When the is evaluated with Opsite Flexigirit, the width of edema increases as the surface width increases. Patients included in the study will be evaluated for approximately 69 days until April 10, 2022.

SECONDARY OUTCOMES:
The effect of the warm wet application on the degree of phlebitis in the care of peripheral intravenous catheter-related phlebitis. | approximately 69 days until 10 April 2022
  The degree of phlebitis before and after the application will be determined according to the phlebitis scale. After the warm wet application, the degree of phlebitis will be determined again and the effectiveness of the warm wet application will be evaluated. The phlebitis scale consists of 5 degrees and as the number of degrees increases, the rate of phlebitis increases. Patients included in the study will be evaluated for approximately 69 days until April 10, 2022.

CONTACTS AND LOCATIONS:
Overall Officials: Fatma Aksoy, RN, Principal Investigator — Ordu University; Sule Bıyık Bayram, PhD, Study Director — Karadeniz Teknik University
Locations (1):
- Fatma Aksoy, Ordu, Turkey (Türkiye)

IPD SHARING:
Plan to Share IPD: No